CLINICAL TRIAL: NCT06724367
Title: TRANSSPINAL DIRECT CURRENT STIMULATION ON FUNCTIONAL MOBILITY IN POST-STROKE PATIENTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 81604324.2.0000.5208
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transspinal direct current stimulation (Experimental): This group will receive 10 sessions of transspinal direct current stimulation associated with gait training.
  Interventions: Device: Transspinal direct current stimulation
- Transspinal direct current stimulation sham (Sham Comparator): This group will receive 10 sessions of sham transspinal direct current stimulation associated with gait training.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Transspinal direct current stimulation — Direct current electrical stimulation applied non-invasively to the spinal cord.
  Arms: Transspinal direct current stimulation
Device: Sham Comparator — transspinal direct current stimulation simulated
  Arms: Transspinal direct current stimulation sham

SUMMARY:
The aim of this clinical trial is to investigate the effects of transspinal direct current stimulation on the functional mobility of post-stroke patients.

The main question it aims to answer is:

Is transspinal direct current stimulation able to improve functional mobility in post-stroke patients?

The researchers will compare transspinal direct current stimulation associated with gait training with sham transspinal direct current stimulation associated with gait training. To verify the effects of stimulation on the functional mobility of post-stroke patients.

Participants:

* They will be assessed before starting the care, after the care has been completed, 15 and 30 days after the care has been completed.
* They will take part in 10 sessions of transspinal direct current stimulation associated with gait training.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischemic or hemorrhagic stroke, provided by a neurologist.
* Age group greater than or equal to 18 years, of both sexes.
* Any stage of the disease.
* Presence of lower limb sensorimotor disorder related to the stroke
* Absence of cognitive impairment verified through the Mini Mental State Examination (score ≥ 18 for illiterate individuals and ≥ 24 for educated individuals) modified for the Brazilian population.

Exclusion Criteria:

* With other neurological injuries
* With vestibular, visual, cardiovascular or osteomyoarticular disorders of the lower limb that may affect the performance of the proposed tests
* Who have a pacemaker or metallic implants in their spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Timed up and go test | From the start of treatment until 30 days after the end of treatment.
  It is an easy-to-use clinical tool that assesses functional mobility. It consists of measuring the time in which an individual is able to get up from a chair, walk for three meters, turn around, go back and sit down again. The test will be carried out three consecutive times, with a 1-minute interval between each attempt, and the value adopted will be the average time (in seconds) taken to carry out the three attempts. It will be measured before starting treatment, immediately afterwards, 15 and 30 days after the end of treatment.

SECONDARY OUTCOMES:
Functional Ambulation Classification | From the start of treatment until 30 days after the end of treatment.
  The Functional Ambulation Classification (FAC) serves as a parameter for monitoring gait progress during rehabilitation, categorically. It also makes it possible to assess the ability to walk for at least three meters on flat and uneven surfaces, as well as analyzing the ability to walk on ramps and up and down steps. The scale is scored from 1 (non-functional) to 6 (independent on level and uneven surfaces), i.e. the higher the score, the better the outcome. It will be measured before starting treatment, immediately afterwards, 15 and 30 days after the end of treatment.
Fugl-Meyer Assessment Scale | From the start of treatment until 30 days after the end of treatment.
  The Fugl-Meyer Assessment Scale is a quantitative instrument used to assess sensorimotor rehabilitation after stroke. Sections E and F, referring to the lower limb, will be used, with a maximum total score of 34 points, and higher scores reflecting better outcomes. It will be measured before starting treatment, immediately afterwards, 15 and 30 days after the end of treatment.
Mini-Balance Evaluation Systems Test (MiniBESTest) | From the start of treatment until 30 days after the end of treatment.
  The Mini-Balance Evaluation Systems Test is a validated scale capable of evaluating balance in patients with neurological disorders. It consists of 14 items and higher scores imply better outcomes. It will be measured before starting treatment, immediately afterwards, 15 and 30 days after the end of treatment.
Modified Ashworth scale | From the start of treatment until 30 days after the end of treatment.
  The modified Ashworth scale is a 6-point ordinal scale that grades the resistance encountered during passive muscle stretching, with higher values representing worse outcomes. It will be applied to the following joints: hip (flexion, extension, abduction and adduction); knee (flexion and extension) and ankle (plantar flexion and dorsiflexion). It will be measured before starting treatment, immediately afterwards, 15 and 30 days after the end of treatment.
Patient Global Impression of Change Scale | Only in the evaluation immediately after treatment.
  The Patient Global Impression of Change Scale is a scale where individuals rate their improvement related to the intervention they have undergone and its score ranges from 1 (no change) to 7 (much better). It will be applied by a researcher not involved in the study, only at the re-evaluation, as it aims to assess the patient perception of improvement after the intervention.

IPD SHARING:
Plan to Share IPD: No